CLINICAL TRIAL: NCT04386499
Title: Effects of Treatment With Resveratrol on Oocyte and Embryo Quality in Patients Undergoing Assisted Reproductive Techniques( ART)
Brief Title: Biological Effects of Treatment With Resveratrol in ART Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Sandro Gerli, Associate Professor of Obstetrics and Gynecology, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR001
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Resveratrol; Folic Acid

STUDY DESIGN:
Intervention Model Description: parallel, single blind, grouped randomised, interventional clinical study
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): A nutraceutical formulation (trade mark Genante) composed of resveratrol, REVIFAST, folic acid, Vitamin D
  Interventions: Dietary Supplement: Resveratrol
- Folic acid (Active Comparator): Folic Acid 400 ug
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Dietary Supplement: Resveratrol — mixture of trans-resveratrol 150 mg (REVIFAST), folic acid 400 mcg, vitamin D, vitamin B12 and vitamin B6
  Other Names: Genante (S&R Farmaceutici S.p.A, Italy)
  Arms: Resveratrol
Dietary Supplement: Folic acid — 400 mcg of folic acid
  Arms: Folic acid

SUMMARY:
To evaluate the effects of a new nutraceutical formulation containing resveratrol (trademark GENANTE) on gamete quality in order to improve the reproductive process during ART.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of a new nutraceutical formulation containing resveratrol (trademark Genante) on gamete quality in order to improve the reproductive protocols during Assisted reproductive technology (ART) protocols.

The study is a randomized, single blind, parallel, comparative, experimental study during the pre-treatment before in vitro fertilization-embryo transfer (IVF-ET). A total number of 100 patients will be enrolled: 50 patients with a pretreatment control group (control group) and 50 patients with experimental pretreatment study group (resveratrol group). Patients will be assigned to groups during the recruitment phase in a randomized manner. In the control group, the treatment will consist of taking 400 microg once a day of folic acid commonly suggested as part of clinical practice, while in the Resveratrol Group, patients will receive one tablet twice a day (two tablets/day) of Genante. It is specified that the pretreatment with Genante includes folic acid in accordance with the clinical practice, 400 total microg per day. Both treatments will last for 3 months before the IVF procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of infertility
* BMI between 18 and 30 kg/m2,
* regular uterine cavity
* normal thyroid function
* normal blood parameters

Exclusion Criteria:

* primary or secondary ovarian failure
* patients who adhered to Bologna Criteria (at least two of the following: advanced maternal age >40, less than 3 oocytes recovered in previous attempts, abnormal ovarian reserve test)
* presence of ovaries inaccessible to the oocyte pick-up,
* persistent ovarian cysts > 20 mm,
* presence of sactosalpinx
* heterologous fertilization, significant systemic disease or other situations unsuitable for ovarian stimulation

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
follicles | 6 months
  Number of follicles >16 mm
oocytes | 6 months
  number of recovered oocytes
MII oocytes | 6 months
  percentage of metaphase II oocytes
fertilization | 6 months
  fertilization rates
embryos | 6 months
  number of embryos
blastocysts | 6 months
  number of blastocysts
gonadotropins days | 6 months
  duration of ovarian stimulation (days)
gonadotropins IU | 6 months
  dosage of gonadotropins (total IU during ovarian stimulation)

SECONDARY OUTCOMES:
embryos number | 18 months
  number of embryos per transfer
implantation | 18 months
  Implantation rate
pregnancy | 18 months
  clinical pregnancy rate
live birth | 18 months
  live birth rate
miscarriage | 18 months
  miscarriage rate

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Gerli, MD, Principal Investigator — University Of Perugia
Locations (1):
- University of Perugia, Piazza Menghini 1, S. Andrea delle Fratte., Perugia, Umbria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerli S, Della Morte C, Ceccobelli M, Mariani M, Favilli A, Leonardi L, Lanti A, Iannitti RG, Fioretti B. Biological and clinical effects of a resveratrol-based multivitamin supplement on intracytoplasmic sperm injection cycles: a single-center, randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Dec;35(25):7640-7648. doi: 10.1080/14767058.2021.1958313. Epub 2021 Aug 1. PMID 34338114